CLINICAL TRIAL: NCT07006363
Title: Investigation of the Immediate Effect of Instrument-Assisted Soft Tissue Mobilization on Hand Reaction Time, Neck Pain and Cervical Joint Position Sense in University Student E-Sports Players: A Single-Blind Randomized Controlled Pilot Study
Brief Title: Investigation of the Immediate Effect of IASTM on Some Parameters in E-Sports Players
Acronym: IASTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Sivas Cumhuriyet Universtiy (Unknown)
Responsible Party: Principal Investigator, Mustafa Oğuz Kethudaoglu, PT, MSc, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IASTM-Esports2025
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cervical Pain, Posterior; Musculoskeletal Disorder of the Neck; Neck Pain; Posture
Keywords: instrument assisted soft tissue mobilization; e-sports; hand reaction time; graston technique; joint position sense; myofascial release; pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After the first evaluation, participants will determine their groups by choosing closed and opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): IASTM: For the application, the participant is seated on a chair, puts his hands together on the bed in front of him and puts his head on his hands (Figure 4). Vaseline cream is applied to the area to be applied to ensure that the Graston Technique instruments slide more easily in the tissue. The application area is the area between the mastoid processes proximally, the acromial processes laterally, and the T2 vertebra level distally. The researcher who will perform the application stands behind the participant. Application is performed for 10 minutes at a 45o angle with 3 different Graston instruments.
  Interventions: Other: IASTM
- Control Group (No Intervention): Members of the Control Group who will not be subjected to the application will be made to wait for 10 minutes (the same duration as the application in the Experimental Group) without doing anything between the two evaluations.

INTERVENTIONS:
Other: IASTM — IASTM: For the application, the participant is seated on a chair, puts his hands together on the bed in front of him and puts his head on his hands (Figure 4). Vaseline cream is applied to the area to be applied to ensure that the Graston Technique instruments slide more easily in the tissue. The application area is the area between the mastoid processes proximally, the acromial processes laterally, and the T2 vertebra level distally. The researcher who will perform the application stands behind the participant. Application is performed for 10 minutes at a 45o angle with 3 different Graston instruments.
  Other Names: Graston Technique; Instrument-Assisted Soft Tissue Mobilization; Myofascial Release
  Arms: Intervention Group

SUMMARY:
Due to the nature of competitive sports, frequent and regular training by e-sports players to increase their performance provides e-athletes with success in the field, but it also increases the time spent in front of the screen. It is known that e-athletes train for an average of 5.5 to 10 hours per day. Therefore, sedentary behavior that develops due to screens is an issue that e-athletes should be careful about. While reasons such as disrupted sleep patterns, increased stress levels and mood changes experienced in the game following increased screen time negatively affect cardiovascular and metabolic health, the fact that e-sports do not require any physical effort also negatively affects the e-sports player's muscular activation. Due to the reasons mentioned, e-sports can cause chronic diseases in the long term. The process from the presence of a stimulus to the execution of the action that will occur following the stimulus is called reaction time. Reaction time can also be described as the value taken when a stimulus exceeds the threshold value, when movement is released or at the beginning of the explosive response. Reaction time consists of stages. The process, which starts with the transmission of the sensory stimulus through the receptors, establishes a perceptual link with the motor response and decides to produce a reactive response, and ends with the process of producing a movement that requires muscular force in the perceptual process. In studies conducted on e-sports players, the most common complaints resulting from long training periods are vision problems and eye fatigue, followed by pain experienced especially in the back, neck and wrist areas. E-sports players perform with poor posture compared to traditional athletes. Games played on mobile phones, especially computer-based games, cause changes in the structure of the spine, pain complaints, movement limitations, and loss of stability and balance. It is argued that the main reason for the pain experienced by approximately half of the players is the anterior displacement of the head due to the prolonged static position spent in front of the screen after a certain number of minutes and the pains brought about by muscle strength imbalances. To our knowledge, there is no study in the literature that investigates the immediate effect of a myofascial release technique applied to university student e-sports players on hand reaction time, neck pain and cervical joint position sense parameters. The aim of this study is to investigate the instantaneous effect of a myofascial release technique, the Graston Technique, on hand reaction time, neck pain and cervical joint position sense in university student e-sports players. Our study is valuable in this respect.

DETAILED DESCRIPTION:
''Electronic sports'' or ''E-sports'' are defined as video games played in a virtual environment in an organized and competitive manner with a specific goal in line with individuals or teams. Although the first steps towards introducing e-sports to the public were taken in the 1970s, it continued to attract attention with the popularity of arcade games in the 1980s. It has also been emphasized that the early 1980s were important years in the history of arcade games. While the first period of e-sports consisted of the times of arcade games, the second period was the period when the use of computers and the internet increased instead of arcade games. It has continued to progress with the variety of games and the variety of internet network technology depending on the developments. E-sports continues to increase its popularity by gaining momentum worldwide with players consisting mainly of the younger population following the development of technology.

Due to the nature of competitive sports, frequent and regular training by e-sports players to increase their performance provides e-sports players with success in the field, but it also increases the time spent in front of the screen. It is known that e-sports players train for an average of 5.5 to 10 hours per day. Therefore, sedentary behavior that develops due to screens is an issue that e-sports players should be careful about. While reasons such as disrupted sleep patterns, increased stress levels and mood changes experienced in the game following increased screen time negatively affect cardiovascular and metabolic health, the fact that e-sports do not require any physical effort also negatively affects the e-sports player's muscular activation. Due to the reasons mentioned, e-sports can cause chronic diseases in the long term.

It is stated that the average career years of a typical professional e-sports players are quite short due to the absolute effort he gives to be the best and to continue in the field. It is expected that this performance of the player, who is expected to make quick and accurate decisions in the moves against the complex visual stimuli presented in the game and the opposing team, will decrease after the age of approximately 24.

The process from the presence of a stimulus to the execution of the action that will occur following the stimulus is called reaction time. Reaction time can also be described as the value taken when a stimulus exceeds the threshold value, when movement is released or at the beginning of the explosive response. Reaction time consists of stages. The process, which starts with the transmission of the sensory stimulus through the receptors, establishes a perceptual link with the motor response and decides to produce a reactive response, and ends with the process of producing a movement that requires muscular force in the perceptual process. Stimuli can be visual, auditory or tactile stimuli. In a study, the reaction time was found to be approximately 190 ms (0.19 sec) for light stimuli and approximately 160 ms (0.16 sec) for sound stimuli. When different studies were examined, the reaction time to visual stimuli was found to be 0.15 s, to auditory stimuli 0.12 - 0.27 s, and to tactile stimuli 0.09 - 0.27 s.

In studies conducted on e-sports players, the most common complaints resulting from long training periods are vision problems and eye fatigue, followed by pain experienced especially in the back, neck and wrist areas. E-sports players perform with poor posture compared to traditional athletes. Games played on mobile phones, especially computer-based games, cause changes in the structure of the spine, pain complaints, movement limitations, and loss of stability and balance. It is argued that the main reason for the pain experienced by approximately half of the players is the anterior displacement of the head due to the prolonged static position spent in front of the screen after a certain number of minutes and the pains brought about by muscle strength imbalances. Professional e-sports players perform up to 400 fine motor movements per minute with minor muscle groups. Clicking/pressing movements originating from controllers used repeatedly for long hours do not remain localized with the fingers and can cause pain or injuries in the hand-wrist, elbow, shoulder and cervical region. Neck pain in particular becomes chronic over time. This is because e-sports players train for long hours and compete in competitions in a bad posture where the head is in an anterior tilt position. There are studies in the literature showing that cervical joint position sense is adversely affected in chronic neck pain.

Since the proprioceptive system provides important informational inputs to the central nervous system for motor planning, a decrease in proprioception may lead to postural changes by causing changes in the control of movement, accuracy and timing of motor commands. Proprioception is necessary for well-adapted sensorimotor control. It plays a role in feedback and feedforward sensorimotor control and muscle stiffness regulation, which are particularly important for movement acuity, joint stability, coordination and balance. Cervical proprioception is uniquely important for head-eye coordination and movement control. Proprioception may be impaired in musculoskeletal disorders due to pain, effusion, trauma and fatigue. There is a strong relationship between cervical disability and neck pain. Among functional changes, active range of motion is an important physical variable for activities of daily living and helps to stabilize and orient the head. In patients with neck pain, it has been proven that the cervical joint range of motion decreases, which may be related to the degree of pain and cervical functionality. In a study, it was shown that the Graston Technique applied to the thoracolumbar fascia increased the range of motion and improved the lumbar joint position sense.

In recent years, the examination and treatment of myofascial pathologies have become an indispensable element of the human neuro-musculoskeletal pathology rehabilitation program. On this basis, many soft tissue techniques and myofascial treatment methods have been developed for a more holistic evaluation and treatment of the human body. Instrument-Assisted Soft Tissue Mobilization (IASTM) is a new range of tools that allow clinicians to efficiently find and treat individuals diagnosed with soft tissue dysfunction. ADYSM is a procedure that has its own indications and limitations, and is rapidly gaining popularity due to its effectiveness and efficiency. Foam Roller, kinesio taping, dry needling, Percussive Massage Technique and Graston Technique applications are some of the IASTM techniques.

One of the most commonly used soft tissue techniques is the Graston Technique, which is a manual therapy approach that uses special instruments to perform static and dynamic soft tissue manipulation, aiming to treat soft tissue limitations and increase tissue flexibility, joint range of motion, and patient functionality. The Graston Technique is a soft tissue mobilization technique performed manually with the help of instruments made of stainless steel. With the Graston Technique, adhesions and limitations in the fascia are eliminated. In this application, the body's self-healing mechanism is used. The tissue healing process is initiated with consciously created microtraumas.

To our knowledge, there is no study in the literature that investigates the immediate effect of a myofascial release technique applied to university student e-sports players on hand reaction time, neck pain and cervical joint position sense parameters. The aim of this study is to investigate the instantaneous effect of a myofascial release technique, the Graston Technique, on hand reaction time, neck pain and cervical joint position sense in university student e-sports players. Our study is valuable in this respect.

ELIGIBILITY:
Inclusion Criteria:

* being a university student
* exercise in front of a screen for at least 3 hours a day
* become a licensed e-sports player
* volunteering to participate in the study

Exclusion Criteria:

* having had upper extremity surgery
* having visual impairment that may affect the research results
* having a neurological problem
* having an orthopedic problem causing neck pain

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Hand Reaction Time | baseline, immediately after the intervention
  In e-sports players, hand reaction speed is a factor that affects their performance. Although there are other methods that evaluate hand reaction time, in this study, since the participants are e-sports players, a mouse and web page based method was preferred ("Aim Trainer" Hand Reaction Time Test). This method tests hand-eye coordination along with hand reaction time. When the test starts, a target board appears on the screen. The participant must point to the target board with the mouse and click 30 times in a row. The average time per target is given in milliseconds as a result of the test.

SECONDARY OUTCOMES:
Neck Pain | baseline, immediately after the intervention
  The level and quality of the cervical region pain felt by the participants will be assessed with the Short Form McGill Pain Questionnaire (SF-MPQ), which has validity and reliability in Turkish. This form provides information about the perceptual, sensory and severity sections in pain perception. The main section of the SF-MPQ includes 15 descriptive adjectives (11 perceptual and 4 sensory) for pain perception. The level of severity felt by the patient is assessed with a numerical value scale (0=none, 1=mild, 2=moderate, 3=severe). In addition, a 10 cm visual analog scale (VAS) is used to measure pain severity. They are asked to indicate the pain they feel during the assessment with an ''X'' mark on the 10 cm scale. According to this scale, a ''0'' value indicates no pain, and a ''10'' value indicates the most severe pain. The distance between the marked point and the starting point is measured. Finally, the patient's total pain intensity is evaluated with a 6-point Likert-type scale
Cervical Joint Position Sense | baseline, immediately after the intervention
  The method described by Revel et al. (1991) will be used in the assessment of cervical joint position sense. In this method, a small laser pointer mounted on a light helmet and a board consisting of circles drawn 1 cm apart from each other are used. The individuals to be assessed are seated in a back-supported chair 90 cm away from the board mounted on the wall. The laser pointer is set to the starting point, the participants' eyes are closed and they are asked to keep this point in their mind. The distance from the laser's final position to the initial position is measured horizontally, vertically and globally in centimeters.
  * Horizontal error: The distance of the point returned after the cervical joint movement to the vertical axis is recorded.
  * Vertical error: The distance of the point returned after the cervical joint movement to the horizontal axis is recorded.
  * Global error: The distance of the point returned after the cervical joint movement to the starting point is record

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Oğuz Kethüdaoğlu, PT, MSc, Principal Investigator — Bahcesehir University, Department of Physiotherapy and Rehabilitation; Sefa Eldemir, PT, PhD, Study Chair — Cumhuriyet University; Ayşenur Canan Benli, PT, MSc, Study Chair — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No